CLINICAL TRIAL: NCT04807166
Title: A Prospective, Single-arm, Multicenter, Exploratory Phase II Study to Evaluate the Efficacy and Safety of Anlotinib Combined With Carboplatin/Paclitaxel as First-line Treatment in Patients With Advanced Ovarian Cancer
Brief Title: Anlotinib Combined With Carboplatin/Paclitaxel as First-line Treatment in Patients With Advanced Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wenjun Cheng (Other)
Responsible Party: Sponsor-Investigator, Wenjun Cheng, Director, Head of Gynecology, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JiangsuCHENG001
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms by Site; Genital Neoplasms, Female; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Carcinoma, Ovarian Epithelial; Ovarian Diseases; Genital Diseases, Female; Endocrine System Diseases; Carcinoma; Anlotinib; Angiogenesis; Antineoplastic Agents; Tyrosine Kinase Inhibitor
Keywords: First-line treatment; Advanced Ovarian Cancer; Anlotinib; Carboplatin/Paclitaxel; Efficacy and Safety
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Neoplasms by Site; Genital Neoplasms, Female; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Carcinoma, Ovarian Epithelial; Ovarian Diseases; Genital Diseases, Female; Endocrine System Diseases; Carcinoma | interventions — anlotinib; CP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Combined With Carboplatin/Paclitaxel (Experimental): Anlotinib Combined With Carboplatin/Paclitaxel
  Interventions: Drug: Drug: Anlotinib; Drug: Drug: Carboplatin/Paclitaxel

INTERVENTIONS:
Drug: Drug: Anlotinib — Anlotinib will be administered orally,once a day (12 mg) on days 1-14 of a 21-day cycle
  Other Names: FOCUS V
Drug: Drug: Carboplatin/Paclitaxel — Paclitaxel 175 mg/m2 was given intravenously for 3 hours, D1 Carboplatin AUC 5 was given intravenously for 1 hour, D1
  Other Names: bobei， Lipusu

SUMMARY:
It has been reported that antiangiogenic drugs combined with chemotherapy as first-line treatment, and subsequent antiangiogenic drugs as maintenance therapy for ovarian cancer can achieve better clinical benefits. Therefore, this study is expected to investigate the efficacy and safety of anlotinib combined with carboplatin/paclitaxel as first-line treatment in patients with advanced ovarian cancer.

DETAILED DESCRIPTION:
This study is a single-arm, multicenter, exploratory phase II study to observe the efficacy and safety of anlotinib combined with carboplatin/paclitaxel as first-line treatment in patients with advanced ovarian cancer. The primary end point are progression free survival; the secondary end points include objective response rate, disease control rate, overall survival and safety. The subjects in this study: patients with newly diagnosed advanced (FIGO stage III-IV) ovarian cancer, including histologically or pathologically confirmed high-grade serous ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be female ≥18 years old;
2. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1；
3. Postoperative administration time: within 12 weeks after the maximum tumor reduction operation;
4. Histologically or pathologically confirmed advanced (FIGO stage III - IV) ovarian cancer, fallopian tube cancer, or primary peritoneal cancer；
5. Subjects have enough organ function: (1) Blood routine(without blood transfusion or hematopoietic stimulating factor within 7 days before screening ): a.Hemoglobin (HB)≥9.0g/L; b.Absolute value of neutrophil (ANC)≥1.5 * 10^9 / L; c.Platelet (PLT)≥80 * 10^9 / L; (2) Liver and Renal function(without blood or albumin transfusion within 7 days before screening ): a. Alanine aminotransferase (ALT) and AST≤2.5 times the upper limit of normal value and ALT (AST≤5 times the upper limit of normal value when liver/bone metastasis) b. total bilirubin ≤1.5 times the upper limit of normal value; c.serum creatinine ≤1.5 times the upper limit of normal value, creatinine clearance≥60 ml/min; (3)Blood coagulation function: a.Activated partial thromboplastin time, international standardized ratio adn prothrombin time ≤1.5 times the upper limit of normal value; b.Doppler echocardiographic evaluation: left ventricular ejection fraction(LVEF)≥ 50%
6. Subjects agreed to join the study and signed informed consent;

Exclusion Criteria:

1. Previously received anti angiogenic drugs including but not limited to small molecules such as anlotinib and apatinib and large molecules such as bevacizumab.

2. Patients allergic to the any test drug.

3. Combined disease/ history:

1. Clinical significant hemoptysis occurred within 3 months before admission (daily hemoptysis was greater than 50ml), or significant clinical bleeding symptoms or definite bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood or above, or suffering from vasculitis, etc;
2. Arteriovenous thrombosis events occurred within 6 months before grouping, such as cerebrovascular accident (including temporary ischemic attack), deep venous thrombosis (except venous thrombosis caused by venous catheterization due to early chemotherapy) and pulmonary embolism;
3. Hypertension, which can not be well controlled by antihypertensive drugs (systolic blood pressure>140 mmHg or diastolic blood pressure>90 mmHg); Myocardial infarction, severe / unstable angina pectoris, cardiac insufficiency above New York Heart Association(NYHA) , supraventricular or ventricular arrhythmias with clinical significance, and symptomatic congestive heart failure occurred within 6 months before grouping;
4. Interstitial lung disease, non-infectious pneumonia or uncontrollable systemic diseases (e.g. diabetes, pulmonary fibrosis and acute pneumonia);
5. Renal insufficiency: urine routine indicates urinary protein ≥ + +, or confirms 24-hour urinary protein ≥ 1.0g;
6. History of live attenuated vaccine vaccination within 28 days before the first study medication or expected live attenuated vaccination during the study period;
7. Human immunodeficiency virus infection or known acquired immunodeficiency syndrome (AIDS); active hepatitis;
8. There were severe infections within 4 weeks before the first administration, including, but not limited to, bacteremia and severe pneumonia requiring hospitalization; active infections requiring systemic antibiotics treatment of grade CTCAE ≥ 2 within 2 weeks before the first administration, or unexplained fever > 38.5 °C during the screening period / before the first administration (the researchers judged that fever caused by tumors could be included in the group); there was evidence of active tuberculosis infection within 1 year before administration;
9. Any other malignant tumor has been diagnosed within 3 years before enrollment, except for fully treated basal cell carcinoma or squamous cell skin cancer or cervical carcinoma in situ;
10. Major surgery was performed within 28 days before enrollment (tissue biopsy required for diagnosis and central venous catheterization via peripheral venipuncture are allowed);
11. Subjects who have previously received or are prepared to receive allogeneic bone marrow transplantation or solid organ transplantation;
12. Patients with peripheral neuropathy ≥2 grade 2; patients with active brain metastasis, carcinomatous meningitis, spinal cord compression, or diseases found in brain or leptomeninges by imaging CT or MRI examination during screening (patients with brain metastasis who had completed treatment 14 days before admission and whose symptoms were stable can be enrolled in the group, but no symptoms of cerebral hemorrhage should be confirmed by cranial MRI, CT or venography)；
13. Factors that significantly affect the absorption of oral drugs, such as inability to swallow, chronic diarrhea, and intestinal obstruction with significant clinical significance

4. Women of child-bearing potential should have negative results of serum or urine pregnancy test. Women must use adequate birth control in the duration of study participation.

5. Other serious physical or mental disorders or laboratory abnormalities that may increase the risk when in this study or interfere with the results of the study, and patients whom the researchers believe are not suitable for this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Through study completion, an average of 1-2 year
  Progression Free Survival (PFS) is defined as the time from the initial treatment to disease progression (defined by RECIST 1.1) or death of any cause

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Through study completion, an average of 1 year
  ORR is defined as the proportion of participants achieving complete response (CR) or partial response (PR) as assessed by RECIST1.1
Disease Control Rate (DCR) | Through study completion, an average of 1 year
  Disease control rate is defined as the proportion of participants achieving complete response (CR), partial response (PR) or stable disease (SD) according to RECIST1.1.
Overall survival (OS) | Through study completion, an average of 1 year
  Overall survival (OS) is defined as time from randomisation to the first occurrence of death from any cause [ Time Frame: From date of treatment beginning until the date of death from any cause
Adverse events (AE) | Through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE 5.0 To further describe safety and assess toxicities encountered with the use of the proposed treatment regimen in participants

CONTACTS AND LOCATIONS:
Overall Officials: Wenjun Cheng, MD,PhD, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (6):
- China (6):
  - Huai'an First People's Hospital, Huai'an
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Affiliated Hospital of Jiangnan University, Wuxi
  - Yancheng No.1 People's Hospital, Yancheng

IPD SHARING:
Plan to Share IPD: No
Contact Prof. Cheng for primary data.